CLINICAL TRIAL: NCT02883868
Title: Stromal Demarcation Line: is it Predictive for Cross-Linking Efficiency?
Acronym: STROMA-CROSS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-09Obs-CHRMT
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-08

CONDITIONS: Progressive Keratoconus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- patients treated with CXL

SUMMARY:
To assess the association between stromal demarcation line after collagen crosslinking (CXL) for progressive keratoconus and mid-term (6 month) refractive, topographic and clinical outcomes of CXL

DETAILED DESCRIPTION:
All consecutive patients treated with CXL between March 2014 and March 2015 were included. They all underwent the same procedure: accelerated-CXL protocol (10 minutes UVA irradiation with 9 mW/cm2 intensity), irradiation device (IROC UV-X™ 2000, Medeuronet). One month after the procedure, AS-OCT examination was performed in all patients (RS-3000, NIDEK). The visibility of the stromal demarcation line was scored (0: not visible line; 1: visible line, but measurement not clearly defined; 2: clearly visible line) and its depth was measured centrally at anytime it was possible. Changes in best corrected visual acuity (BCVA), spherical equivalent (SE), Kmax and thinnest pachymetry, were studied preoperatively and at 6 months

ELIGIBILITY:
Inclusion Criteria:

* patients treated with CXL

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients treated with CXL between March 2014 and March 2015 were included
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
visibility of the stromal demarcation line | month 1